CLINICAL TRIAL: NCT00408889
Title: Prospective Evaluation of Predictors for Organ Failure Following Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Other Study IDs: post OLT
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Last update posted 2010-04-09 (Estimated); Status verified 2008-12

CONDITIONS: Liver Transplantation
Keywords: liver transplantation; organ failure; outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Early organ failure occurs frequently and is difficult to predict. The study aims to define a predictive score for early transplant failure.

DETAILED DESCRIPTION:
Patients will be monitored 7 days following liver transplantation, including clinical scores, clinical chemistry, ultrasound findings and indocyaninegreen-clearance.

ELIGIBILITY:
Inclusion Criteria:

* orthotopic liver transplantation
* age > 18 years

Exclusion Criteria:

* allergy to indocyangreen

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Eisenbach, Dr., Principal Investigator — Heidelberg University
Locations (1):
- University Hospital of Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Schneider L, Spiegel M, Latanowicz S, Weigand MA, Schmidt J, Werner J, Stremmel W, Eisenbach C. Noninvasive indocyanine green plasma disappearance rate predicts early complications, graft failure or death after liver transplantation. Hepatobiliary Pancreat Dis Int. 2011 Aug;10(4):362-8. doi: 10.1016/s1499-3872(11)60061-1. PMID 21813383